CLINICAL TRIAL: NCT06993571
Title: Closed-loop Phase-adaptive Cerebellar Transcranial Alternating Current Stimulation (tACS) to Modulate Activity in the Cerebello-thalamo-cortical Network to Reduce Parkinson's Disease Tremor
Brief Title: Cerebellar Transcranial Alternating Current Stimulation (tACS) to Modulate Parkinson's Disease Tremor
Acronym: tACS_PD_TR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Simone Zittel, Dr. med., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Cereb_tACS_PD_TR
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease (PD); Tremor
Keywords: Parkinson's disease; Hand tremor; Transcranial alternating current stimulation; Non-invasive brain stimulation; Closed-loop stimulation; Phase-adaptive stimulation; Tremor entrainment
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Intervention Model Description: Each participant will receive active, sham, and control stimulation in a randomized manner.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active-tACS (Experimental): Patients receive an active tACS stimulation with 2-4 mA amplitude
  Interventions: Device: Active-tACS
- Sham-tACS (Sham Comparator): Patients receive a tACS stimulation with 0 mA amplitude
  Interventions: Device: Sham-tACS
- Unlocked-tACS (Active Comparator): Patients receive an active tACS stimulation with 2-4 mA amplitude but without phase alignment between tremor and tACS
  Interventions: Device: Unlocked-tACS

INTERVENTIONS:
Device: Active-tACS — 30 seconds of closed-loop tACS at 2-4 mA, with 6 alternating phase alignments and 1-3 repetitions. Phase alignment is adjusted to the patient's tremor frequency and rhythm in real time. Administered using the neuroConn LOOPIT device and 2 electrodes placed on the cerebellum and jaw, with an area of 5x5 and 5x7 respectively. The stimulation begins with a 3-second ramp-up and ends with a 3-second ramp-down.
  Arms: Active-tACS
Device: Sham-tACS — 30 seconds of tACS at 0 mA and 1-3 repetitions. Administered using the neuroConn LOOPIT device and 2 electrodes placed on the cerebellum and jaw, with an area of 5x5 and 5x7 respectively. The sham protocol begins with a 3-second ramp-up and ends with a 3-second ramp-down.
  Arms: Sham-tACS
Device: Unlocked-tACS — 30 seconds of open-loop tACS at 2-4 mA, with no phase alignments and 1-3 repetitions. Administered using the neuroConn LOOPIT device and 2 electrodes placed on the cerebellum and jaw, with an area of 5x5 and 5x7 respectively. The stimulation begins with a 3-second ramp-up and ends with a 3-second ramp-down.
  Arms: Unlocked-tACS

SUMMARY:
Parkinson's disease (PD) is a prevalent neurodegenerative disorder characterized by different motor symptoms, including tremor, which is particularly difficult to manage. Common treatments, such as dopaminergic therapy, can have limitations in efficacy. Recent advancements in non-invasive brain stimulation, specifically phase-adaptive transcranial alternating current stimulation (tACS), offer a promising approach to reduce PD tremor. In the current project, a newly developed closed-loop system delivers precisely synchronized cerebellar tACS by aligning stimulation with the intrinsic hand tremor signal. The study will assess the efficacy of this novel approach to reduce hand tremor in PD patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder, characterized by progressive neurodegeneration, especially in the substantia nigra. Clinically, PD is characterized by motor impairment, including bradykinesia, rigidity, postural instability, and tremor, with hand trem-or being particularly challenging due to its heterogeneity and the incomplete understanding of its underlying neurophysiological mechanisms. Emerging evidence suggests that pathological activity in the cortico-thalamo-cortical (CTC) network is associated with PD tremor amplitude. In recent years, the cerebellum has been recognized for its direct involvement in tremor dynamics within the CTC network. Addressing the abnormal oscillatory activity within this network could potentially modu-late tremor pathophysiology.

Current therapeutic approaches for PD tremor focus on dopaminergic replacement, however some patients exhibit minimal response to this treatment. Deep brain stimulation (DBS) has shown effi-cacy in alleviating tremor, but its invasive nature and associated risks limit its widespread use. Con-sequently, there has been growing interest in non-invasive brain stimulation techniques as poten-tial alternatives for tremor management. Among these techniques, transcranial alternating current stimulation (tACS) has gained significant attention due to its ability to modulate endogenous brain oscillations. Phase-specific tACS, which involves aligning the stimulation phase with the intrinsic tremor rhythms, has demonstrated potential in entraining and reducing PD tremor. However, the application of this technique has been constrained by the complexities associated with phase ad-justment algorithms and the need for a responsive closed-loop system capable of real-time phase synchronization.

For the current project, a novel closed-loop device has been developed together with the collabo-rator neuroConn GmbH that is specifically designed to target PD tremor. This device is capable of real-time monitoring of hand tremor, rapid signal processing, and delivering phase-locked tACS within safe operational parameters. The central hypothesis is that phase-locked tACS of the cere-bellum can modulate the oscillatory dynamics within the CTC network and thereby reduce tremor amplitude in PD patients.

The study will involve PD patients with moderate to severe hand tremor, as assessed using the Movement Disorders Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The experimental design involves two sessions, both utilizing closed-loop tACS at an intensity of 2 to 4 mA.

In each session, a baseline recording of PD hand tremor will be collected before stimulation. In the first session, the phase alignment between the tremor and tACS signals will be systematically varied across 60° phase bins; plus a sham (zero stimulation amplitude) and an unlocked stimulation proto-col (open-loop). The data from this session will be analyzed to determine the optimal phase align-ment. In the second session, tACS will be applied using the optimal phase alignment identified in the first session. After each block of stimulation, a post-stimulation baseline recording will be con-ducted to evaluate the immediate effects of the intervention. This design enables the assessment of phase-specific effects of closed-loop tACS on PD hand tremor.

This study aims to assess the extent and duration of tremor reduction achieved by closed-loop phase-adaptive cerebellar tACS, enhancing our understanding of the CTC network and potentially offering new insights into non-invasive therapeutic strategies for managing PD tremor.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease based on UK Brain Bank criteria
* Patient exhibiting moderate to severe hand tremor
* Provision written informed consent by the patient

Exclusion Criteria:

* History of other neurological disorders such as vascular malformations, ischemic or haemorrhagic stroke, cerebral neoplasia, epilepsy, or major psychiatric illness
* Existence of heart pacemaker or metal implants in the body
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tremor reduction | During the stimulation
  A significant reduction in the amplitude of hand tremor as the active tACS stimulation with the optimum phase alignment is being delivered. Tremor amplitude is computed offline in MATLAB.

SECONDARY OUTCOMES:
Tremor entrainment | During the stimulation
  Changes in tremor characteristics including instantaneous frequency due to active stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Due to data protection policies